CLINICAL TRIAL: NCT07134556
Title: A Phase II Trial Evaluating the Safety and Efficacy of the Combination of Zimberelimab, Domvanalimab and Sacituzumab Govitecan as First-line Therapy for PD-L1 Positive Advanced Triple-negative Breast Cancer
Brief Title: Phase II Trial Evaluating the Safety and Efficacy of the Combination of Zimberelimab, Domvanalimab and Sacituzumab Govitecan as 1L Therapy for PD-L1 Positive Advanced TNBC
Acronym: ADJUNCT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDOPP0653; 2025-521489-80 (EudraCT Number)
Record Dates: First submitted 2025-08-06; First posted 2025-08-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-08

CONDITIONS: Triple Negative Breast Cancer; PDL-1 Positive
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — zimberelimab; sacituzumab govitecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- zimberelimab, domvanalimab and sacituzumab govitecan (Experimental): patients will receive zimberelimab as an intravenous infusion (IV) at a dose of 360 mg on Day 1 (D1); domvanalimab as an IV at a dose of 1200 mg on D1 and sacituzumab govitecan as an IV at a dose of 10 mg/kg on D1 and 8 D8 of each 21-day cycle until unacceptable toxicity, disease progression, death, discontinuation from the Study treatment for any other reason or End of Study (EoS), whichever occurs first.
  Interventions: Drug: Zimberelimab (AB122); Drug: Domvanalimab (DOM); Drug: Sacituzumab Govitecan (SG)

INTERVENTIONS:
Drug: Zimberelimab (AB122) — Patients will receive zimberelimab as an IV at a dose of 360 mg on D1 of each 21-day cycle until unacceptable toxicity, disease progression, death, discontinuation from the Study treatment for any other reason or End of Study (EoS), whichever occurs first.
Drug: Domvanalimab (DOM) — Patients will receive domvanalimab as an IV at a dose of 1200 mg on D1 of each 21-day cycle until unacceptable toxicity, disease progression, death, discontinuation from the Study treatment for any other reason or End of Study (EoS), whichever occurs first.
Drug: Sacituzumab Govitecan (SG) — Patients will receive sacituzumab govitecan as an IV at a dose of 10 mg/kg on D1 and D8 of each 21-day cycle until unacceptable toxicity, disease progression, death, discontinuation from the Study treatment for any other reason or End of Study (EoS), whichever occurs first.

SUMMARY:
The ADJUNCT is a single-arm, phase II clinical trial to evaluate the safety and efficacy of the combination of zimberelimab, domvanalimab and sacituzumab govitecan as first-line therapy for patients with PD-L1 positive advanced or metastatic triple-negative breast cancer.

DETAILED DESCRIPTION:
This is a single-arm, phase II clinical trial to evaluate the safety and efficacy of the combination of zimberelimab, domvanalimab and sacituzumab govitecan as first-line therapy for patients with PD-L1 positive advanced or metastatic triple-negative breast cancer. Patients ≥18 years with PD-L1 positive (Combined Positive Score [CPS] ≥10, assessed using the PD-L1 IHC 22C3 pharmDx assay) advanced TNBC that is not amenable to treatment with curative intent, who have measurable disease and have not received prior systemic treatment in the advance setting. Patients who have received prior (neo)adjuvant therapies are permitted if the disease-free interval (DFI) is at least 6 months.

Evidence of measurable disease as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v.1.1), Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, and adequate bone marrow and organ function are mandatory.

Patients will receive zimberelimab as an intravenous infusion (IV) at a dose of 360 mg on Day 1; domvanalimab as an IV at a dose of 1200 mg on Day 1 and sacituzumab govitecan as an IV at a dose of 10 mg/kg on Days 1 and 8 of each 21-day cycle until unacceptable toxicity, disease progression, death, discontinuation from the Study treatment for any other reason or End of Study (EoS), whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male participants, regardless of race and/or ethnic group, aged 18 years or older, able to understand and give written informed consent form (ICF).
2. Histologically confirmed TNBC per American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) 2018 criteria, based on local testing performed on the most recent biopsy in the metastatic setting. . Triple-negative status is defined as <1% expression for estrogen receptor (ER) and progesterone receptor (PgR) and negative for human epidermal growth factor receptor 2 (HER2) (0-1+ by immunohistochemistry or 2+ and negative by in situ hybridization test).
3. PD-L1 positive status defined as a CPS ≥ 10 determined by the antibody 22C3 PharmDx assay, based on local testing.
4. Unresectable locally advanced or metastatic disease documented by computerized tomography (CT) scan or magnetic resonance imaging (MRI) that is not amenable to resection with curative intent.
5. Measurable disease according to RECIST v.1.1. Tumor lesions situated in a previously irradiated area are considered measurable if unequivocal progression has been documented in such lesions since radiation.
6. No prior systemic therapy for advanced disease. For patients receiving (neo)adjuvant therapy, a disease-free interval of at least 6 months between completion of systemic treatment with curative intent and first documented local or distant disease recurrence is mandatory. Dates of postoperative radiotherapy are not included in this calculation. Prior use of an anti-PD-L1 agent in the curative TNBC setting is permitted.
7. Have adequate bone marrow, liver, and renal function.
8. Resolution of all acute toxic effects of previously administered agent to grade ≤ 1 as determined by the US National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (v.5.0) (except for alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion).
9. Willingness and ability to provide the most recently available formalin-fixed paraffin-embedded (FFPE) tumor tissue sample from the metastatic site at the time of inclusion. If this archival tissue is not available, a newly obtained baseline biopsy of an accessible tumor lesion is required before the start of Study treatment. If obtaining a biopsy is not feasible, patient eligibility must be evaluated by the Medical Monitor.
10. Willingness to provide blood and stool samples at the established time points.
11. Women of childbearing potential who are sexually active with a non-sterilized male partner must have a negative serum pregnancy test within 14 days before Study treatment initiation. In addition, they must agree to use one highly effective method of birth control from the time of screening until 6 months after the last dose of Study treatments. Female patients must refrain from egg cell donation and breastfeeding during this same period.
12. Male participants who are sexually active with a female partner of childbearing potential must be surgically sterile or using an acceptable method of contraception from the time of screening until 6 months after the last administration of the Study drug. Male participants must not donate or bank sperm during this same period.
13. ECOG performance status of 0-1.
14. Minimum life expectancy of ≥ 12 weeks at screening.

Exclusion Criteria:

1. Inability to comply with Study and follow-up procedures.
2. Pregnant or lactating women or patients not willing to apply highly effective contraception as defined in the protocol.
3. Concomitant participation in a Study with an investigational agent or investigational device within 4 weeks prior to Study enrolment. Participants enrolling in observational studies are eligible.
4. Have previously been treated with chemotherapy or immunotherapy in the metastatic setting.
5. Have previously been treated with topoisomerase 1 inhibitors or antibody drug conjugates containing a topoisomerase inhibitor in the curative setting.
6. Have known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases (except those treated with chemotherapy) may participate if they meet the following criteria: stable CNS disease demonstrated by radiographic stability for at least 4 weeks prior to enrollment, all neurologic symptoms have returned to baseline, no evidence of new or enlarging brain metastases, and clinical stability for at least 2 weeks while taking ≤ 10 mg/day of prednisone or its equivalent. However, all participants with carcinomatous meningitis are excluded regardless of clinical stability.
7. Have a concurrent malignancy or malignancy within 3 years of Study enrollment except for participants with surgically cured carcinoma in situ of the cervix, non-melanoma skin carcinoma, or stage I uterine cancer, that are allowed to enroll. For other cancers considered to have a low risk of recurrence, discussion with the Sponsor's Medical Monitor is required.
8. Known allergy or hypersensitivity reaction to any investigational medicinal product (IMP) including zimberelimab, sacituzumab govitecan and domvanalimab or any of their components.
9. Requirement for ongoing therapy with any prohibited medications listed in the protocol.
10. Have received prior radiotherapy within 2 weeks of start of Study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A two-week washout period is permitted for palliative radiation to non-CNS disease.
11. Major surgical procedure or significant traumatic injury within 14 days before the first dose of Study treatment or anticipation of need for major surgery within the course of the Study treatment.
12. Have active chronic inflammatory bowel disease (ulcerative colitis/Crohn's disease) or gastrointestinal perforation within 6 months of enrollment.
13. Have an active cardiac disease or a history of cardiac dysfunction or conduction abnormalities.
14. Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (e.g., pulmonary emboli within three months of the Study enrolment, severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disease, pleural effusion, post COVID-19 pulmonary fibrosis, etc.), and any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement (e.g., rheumatoid arthritis, Sjogren's syndrome, sarcoidosis, etc.), or prior pneumonectomy.
15. Have a history of non-infectious interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
16. Have an active autoimmune disease that has required systemic treatment in the past 2 years (e.g., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs) or are receiving chronic systemic corticosteroids at doses > 10 mg/day prednisone or its equivalent 4 weeks prior to the first dose of study drug. Use of topical, inhalational, intranasal, and intraocular steroids and use as premedication for known hypersensitivity reactions (eg, intravenous [IV] contrast, IV drug infusions) will be permitted. Replacement therapy (e.g., thyroxine, insulin, physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed. Additionally, patients who have experienced immune-related adverse events (irAEs) due to prior early-stage PD-L1 treatment and for whom rechallenge with a PD-L1 drug may pose a risk should also be excluded.
17. Current known infection with hepatitis B virus (HBV), or hepatitis C virus (HCV). Patients with past HBV infection or resolved HBV infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive hepatitis B core antibody [HBcAb] test, accompanied by a negative HBV DNA test) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
18. Have uncontrolled primary immunodeficiency, known human immunodeficiency virus (HIV) infection.
19. Other active uncontrolled infection at the time of enrollment.
20. Have undergone an allogenic tissue or solid organ transplant.
21. Receipt of live or attenuated vaccine within 30 days prior to the first dose of Study treatment.
22. A history of uncontrolled seizures, central nervous system (CNS) disorders, or serious and/or unstable pre-existing psychiatric disability judged by the investigator to be clinically significant and adversely affecting compliance to Study drugs or interfering with subject safety.
23. Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the Study.
24. Known substance abuse or any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate patient participation.
25. Inability or unwillingness to comply with the requirements of the protocol in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-05-28 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
Efficacy in terms of objective response rate (ORR) as per RECIST v.1.1. | Approximately 1 year
  ORR rate defined as the rate of patients with complete response (CR) or partial response (PR) as determined locally by the investigator in accordance RECIST v.1.1.

SECONDARY OUTCOMES:
Efficacy in terms of PFS as per RECIST v.1.1. | Aproximately 1 year
  PFS: period from treatment initiation until the first occurrence of disease progression as determined locally by the investigator assessment using RECIST v.1.1 or death from any cause, whichever occurs first.
Efficacy in terms of Overall Survival. | Aproximately 1 year
  OS: period from treatment initiation until death from any cause.
Efficacy in terms of Clinical benefit rate (CBR) as per RECIST v.1.1. | Aproximately 1 year
  CBR: rate of patients with objective response (CR or PR), or stable disease for at least 24 weeks, as determined locally by the investigator using RECIST v.1.1.
Efficacy in terms of Time to response (TTR) as per RECIST v.1.1. | Aproximately 1 year
  TTR: period from treatment initiation to the first objective tumor response (tumor shrinkage of ≥ 30%) observed for patients who achieved a CR or PR, as determined locally by the investigator using RECIST v.1.1.
Efficacy in terms of Duration of response (DoR) as per RECIST v.1.1. | Aproximately 1 year
  DoR: period from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first, as determined locally by the investigator using RECIST v.1.1.
Efficacy in terms of Best percentage of change as per RECIST v.1.1. | Aproximately 1 year
  Best percentage of change from baseline in the size of target tumor lesions, defined as the biggest decrease, or smallest increase if no decrease will be observed, as determined locally by the investigator using RECIST v.1.1.
To evaluate changes in health-related quality-of-life (QoL) | Approximately 1 year
  Changes from baseline in the European Organization for Research and Treatment of Cancer (QoL) Questionnaire Core 30 (EORTC QLQ-C30) scale.
  The EORTC-QLQ-C30 is a 30-item questionnaire, composed of five multi-item functional subscales (physical, role, emotional, cognitive, and social functioning), three multi-item symptom scales (fatigue, nausea/vomiting, and pain), a global QoL subscale, and six single-item symptom scales assessing other cancer-related symptoms (dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and the financial impact of cancer). The questionnaire employs 28 4-point Likert scales with responses from "not at all" to "very much" and two 7-point Likert scales for global health and overall QoL. Responses to all items are then converted to a 0 to 100 scale. For functional and global QoL scales, higher scores represent a better level of functioning/QoL. For symptom-oriented scales, a higher score represents more severe symptoms.
To evaluate changes in health-related quality-of-life (QoL) | Approximately 1 year.
  Changes from baseline in the European Organization for Research and Treatment of Cancer (QoL) Questionnaire BR42 (QLQ-BR42).
  The EORTC-QLQ-BR42 is a 42-item BC-specific companion module to the EORTCQLQ-C30 and consists of nine multi-item scales that assess body image, sexual functioning, breast satisfaction, systemic therapy side effects, arm symptoms, breast symptoms, endocrine therapy symptoms, skin mucosis symptoms, endocrine sexual symptoms; single items assess sexual enjoyment, future perspective, and feelings about upset by hair loss.
To determine the safety and toxicity profile of zimberelimab, sacituzumab govitecan and domvalimab treatment. | Approximately 1 year
  Safety and tolerability as per NCI-CTCAE v.5.0. Safety assessments will consist of monitoring and recording protocol-defined AEs, SAEs and non-serious adverse event of special interests (AESIs); measurement of protocol-specified hematology, clinical chemistry, measurement of protocol-specified vital signs; and other protocol specified tests that are deemed critical to the safety evaluation of the Study drug(s).

CONTACTS AND LOCATIONS:
Overall Officials: Tim Robinson, BMBS, PhD, Principal Investigator — University of Bristol, Bristol, England (UK)

IPD SHARING:
Plan to Share IPD: No